CLINICAL TRIAL: NCT04958005
Title: Evaluation of Salivary Interleukin-32, Interleukin-10, Interleukin-6 and Tumor Necrosis Factor-alpha Levels in Children With Early Childhood Caries.
Brief Title: Salivary Interleukin-32, Interleukin-10, Interleukin-6 and Tumor Necrosis Factor-alpha Levels in Children
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Sultan KELES, Assoc.Prof.Dr., Aydin Adnan Menderes University
Other Study IDs: 2020/190
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Early Childhood Caries
Keywords: early childhood caries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with early chilhood caries: Early chilhood caries group
  Interventions: Diagnostic Test: ELISA
- Without early chilhood caries: Control group
  Interventions: Diagnostic Test: ELISA

INTERVENTIONS:
Diagnostic Test: ELISA — Enzim linked immunoabsorbant assay

SUMMARY:
This study aimed to evaluate the levels of interleukin 10, interleukin 6, interleukin 32 and tumor necrosis factor-alpha (TNF-α) in saliva of children with early childhood caries.

DETAILED DESCRIPTION:
Fifty six children ( 28 with early childhood caries and 28 without early childhood caries ; age range 3-6 years) will be recruited for the study. Probing pocket depth (PPD), gingival index (GI) and plaque index (PI) will be recorded and saliva samples will be collected. Interleukin-32, Interleukin-10, Interleukin-6 and TNF-α will be analyzed in saliva samples by ELISA.

ELIGIBILITY:
Inclusion Criteria:

* Children with untreated early chilhood caries
* Age between 3 and 6 years

Exclusion Criteria:

* Having a systemic problem or mental retardation
* Children with treated caries

Ages: 3 Years to 70 Months | Sex: All
Age Groups: Child
Study Population: 28 children with early childhood caries and 28 children without caries will be collected.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
IL-32 | Baseline
  Interleukin- 32 level
IL-10 | Baseline
  Interleukin- 10 level

SECONDARY OUTCOMES:
IL-6 | Baseline
  Interleukin- 6 level
Tnf-Alpha | Baseline
  Tnf-alpha level

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan KELEŞ, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided